CLINICAL TRIAL: NCT04023045
Title: Evaluation of an Energy-Harvesting Knee Prosthesis in Transfemoral Prosthesis Users
Brief Title: Assist-Knee: Energy-Harvesting Knee Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthocare Innovations, LLC (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 7826-01; 1R43HD097826 (NIH)
Record Dates: First submitted 2019-06-27; First posted 2019-07-17 (Actual); Results first posted 2022-10-07 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Transfemoral Amputation; Artificial Limbs

STUDY DESIGN:
Intervention Model Description: Crossover clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Habitual Prosthesis (Active Comparator): Participant's prescribed prosthesis
  Interventions: Device: Habitual Prosthesis
- Assist-Knee (Experimental): Experimental knee prosthesis
  Interventions: Device: Assist-Knee

INTERVENTIONS:
Device: Assist-Knee — Assist-Knee is an experimental lower limb knee prosthesis.
  Arms: Assist-Knee
Device: Habitual Prosthesis — Habitual baseline prosthesis prescribed by participant's clinician.
  Arms: Habitual Prosthesis

SUMMARY:
The purpose of this research is to validate the Assist-Knee design and function by collecting pilot data during the stand-to-sit-to-stand transition in transfemoral prosthesis users when using the Assist-Knee to harvest energy and return energy .

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transfemoral limb loss
* At least one year post-amputation and currently successfully using a prosthesis
* Uses modular endoskeletal prosthetic components
* Has bilateral normal range of motion
* Ability to perform the following activities:
* Walking ability or ability to take steps over 10 meters
* Upright standing stability
* Stand-to-sit stability (i.e. go from a standing position to a seated position independently)
* Sit-to-stand stability (i.e. rise from a seated position independently)
* Ability to communicate individual perceptions in the English language
* Ability to provide informed consent

Exclusion Criteria:

* Confounding injury or musculoskeletal problem
* Pregnancy
* Lower limb peripheral neuropathy
* Symptomatic cardiovascular disease or chronic obstructive pulmonary disease
* Not able to read and understand English
* Use of assistive devices for sit-to-stand and stand-to-sit (e.g. canes, walkers)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Chang, PhD, Principal Investigator — Orthocare Innovations, LLC
Locations (1):
- Orthocare Innovations, LLC, Edmonds, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals were recruited from a sample of convenience in the local area between 07/15/2019 and 02/26/2020.
Groups:
- Assist-Knee (Settings 1): Experimental knee prosthesis
  Assist-Knee: Assist-Knee is an experimental lower limb knee prosthesis. Settings 1: First set of settings tested on Assist-Knee with the participant.
- Assist-Knee (Settings 2): Experimental knee prosthesis
  Assist-Knee: Assist-Knee is an experimental lower limb knee prosthesis. Settings 2: Second set of settings tested on Assist-Knee with the participant.
Period: Habitual Prosthesis Condition
Arm/Group | Habitual Prosthesis | Assist-Knee (Settings 1) | Assist-Knee (Settings 2)
Started | 3 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Assist-Knee (Settings 1) Condition
Arm/Group | Habitual Prosthesis | Assist-Knee (Settings 1) | Assist-Knee (Settings 2)
Started | 0 | 3 | 0
Completed | 0 | 3 | 0
Not Completed | 0 | 0 | 0
Period: Assist-Knee (Settings 2) Condition
Arm/Group | Habitual Prosthesis | Assist-Knee (Settings 1) | Assist-Knee (Settings 2)
Started | 0 | 0 | 3
Completed | 0 | 0 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Participants: Study participants completed both arms of the study: Habitual and Assist-Knee.
  Habitual Prosthesis: Habitual baseline prosthesis prescribed by participant's clinician.
  Assist-Knee Prosthesis: Assist-Knee is an experimental lower limb knee prosthesis.
Arm/Group | Study Participants
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Sit-to-Stand
Description: The amount of time, measured in seconds, needed by the subject to complete the sit-to-stand transition. At least four trials of the sit-to-stand maneuver were collected for each participant using a motion analysis system. Average and standard deviation of the time to complete the sit-to-stand transition were calculated for each participant (each participant served as their own control in this pilot study). The start of the transition was determined by participant initiation; the end of the transition was determined by the participant reaching full knee extension.
Time Frame: Collection at baseline
Population: Each participant served as their own control in this analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Habitual Prosthesis
Number analyzed (Participants) | 3
seconds
  Participant A: number analyzed (Participants) | 1
  Participant A | 1.6 (0.1)
  Participant B: number analyzed (Participants) | 1
  Participant B | 2.2 (0.2)
  Participant C: number analyzed (Participants) | 1
  Participant C | 1.4 (0.2)
Statistical Analysis 1: Comparison: Habitual Prosthesis; Test type: Other; Descriptive analyses (mean and standard deviation) were used to compare the Habitual condition to the Assist-Knee conditions

2. Primary Outcome: Time to Complete Sit-to-Stand
Description: as for outcome 1
Time Frame: After acclimation to Assist-Knee (Participants are given at least 10 minutes and no more than 60 minutes to acclimate to each Assist-Knee condition for safety. After acclimating, participants will complete the maneuver to measure this outcome.)
Population: Each participant served as their own control in this analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Assist-Knee (Settings 1) | Assist-Knee (Settings 2)
Number analyzed (Participants) | 3 | 3
seconds
  Participant A: number analyzed (Participants) | 1 | 1
  Participant A | 3.4 (0.6) | 2.7 (0.2)
  Participant B: number analyzed (Participants) | 1 | 1
  Participant B | 6.4 (1.3) | 3.8 (0.5)
  Participant C: number analyzed (Participants) | 1 | 1
  Participant C | 2.4 (0.5) | 2.9 (0.5)
Statistical Analysis 1: Comparison: Assist-Knee (Settings 1) vs Assist-Knee (Settings 2); Test type: Other; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Timed Up and Go (TUG) Test
Description: The Timed Up and Go (TUG) test is a validated timed functional test that involves standing up from a chair, walking forward for 3 meters, turning around, walking back to the chair for 3 meter, and sitting down. Each participant completed the TUG test for three trials. Time was measured using a stopwatch. Average and standard deviation of the time to complete the TUG test were calculated for each participant (each participant served as their own control in this pilot study).
Time Frame: Collection at baseline
Population: Each participant served as their own control in this analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Habitual Prosthesis
Number analyzed (Participants) | 3
seconds
  Participant A: number analyzed (Participants) | 1
  Participant A | 7.1 (0.5)
  Participant B: number analyzed (Participants) | 1
  Participant B | 13.7 (1.0)
  Participant C: number analyzed (Participants) | 1
  Participant C | 12.3 (0.8)
Statistical Analysis 1: Comparison: Habitual Prosthesis; Test type: Other; [other analysis details as in outcome 1, analysis 1]

4. Secondary Outcome: Timed Up and Go (TUG) Test
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Each participant served as their own control in this analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Assist-Knee (Settings 1) | Assist-Knee (Settings 2)
Number analyzed (Participants) | 3 | 3
seconds
  Participant A: number analyzed (Participants) | 1 | 1
  Participant A | 12.3 (1.1) | 12.8 (0.8)
  Participant B: number analyzed (Participants) | 1 | 1
  Participant B | 25.0 (3.0) | 22.0 (1.4)
  Participant C: number analyzed (Participants) | 1 | 1
  Participant C | 20.8 (3.5) | 18.8 (1.5)
Statistical Analysis 1: Comparison: Assist-Knee (Settings 1) vs Assist-Knee (Settings 2); Test type: Other; [other analysis details as in outcome 1, analysis 1]

5. Secondary Outcome: Time to Complete Stand-to-Sit
Description: The amount of time, measured in seconds, needed by the subject to complete the stand-to-sit transition. At least four trials of the stand-to-sit maneuver were collected for each participant using a motion analysis system. Average and standard deviation of the time to complete the stand-to-sit transition were calculated for each participant (each participant served as their own control in this pilot study). The start of the transition was determined by participant initiation; the end of the transition was determined by the participant being seated on a chair.
Time Frame: Collection at baseline
Population: Each participant served as their own control in this analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Habitual Prosthesis
Number analyzed (Participants) | 3
seconds
  Participant A: number analyzed (Participants) | 1
  Participant A | 2.7 (0.1)
  Participant B: number analyzed (Participants) | 1
  Participant B | 4.1 (1.0)
  Participant C: number analyzed (Participants) | 1
  Participant C | 1.6 (0.2)
Statistical Analysis 1: Comparison: Habitual Prosthesis; Test type: Other; [other analysis details as in outcome 1, analysis 1]

6. Secondary Outcome: Time to Complete Stand-to-Sit
Description: as for outcome 5
Time Frame: as for outcome 2
Population: Each participant served as their own control in this analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Assist-Knee (Settings 1) | Assist-Knee (Settings 2)
Number analyzed (Participants) | 3 | 3
seconds
  Participant A: number analyzed (Participants) | 1 | 1
  Participant A | 4.4 (0.4) | 3.3 (0.4)
  Participant B: number analyzed (Participants) | 1 | 1
  Participant B | 4.9 (1.7) | 4.5 (0.9)
  Participant C: number analyzed (Participants) | 1 | 1
  Participant C | 2.5 (0.1) | 2.7 (0.7)
Statistical Analysis 1: Comparison: Assist-Knee (Settings 1) vs Assist-Knee (Settings 2); Test type: Other; [other analysis details as in outcome 1, analysis 1]

7. Secondary Outcome: Percentage of Body Weight on Contralateral Limb at 65 Degrees Knee Flexion
Description: The percentage of body weight on the contralateral limb was determined for both stand-to-sit and sit-to-stand transitions at 65 degrees knee flexion. A force plate under the contralateral limb recorded the amount of loading on the limb during the stand-to-sit and sit-to-stand transitions. The amount of contralateral limb loading at 65 degrees knee flexion was determined and divided by the participant's total loading due to overall body weight. This value was then converted to a percentage.
Time Frame: Collection at baseline
Population: Each participant served as their own control in this analysis.
Measure: Mean (Standard Deviation); unit: % body weight
Groups:
- SIT With Habitual Prosthesis: Contralateral limb weight distribution during stand-to-sit at 65 degrees knee flexion when using habitual prosthesis.
- STAND With Habitual Prosthesis: Contralateral limb weight distribution during sit-to-stand at 65 degrees knee flexion when using habitual prosthesis.
Arm/Group | SIT With Habitual Prosthesis | STAND With Habitual Prosthesis
Number analyzed (Participants) | 3 | 3
% body weight
  Participant A: number analyzed (Participants) | 1 | 1
  Participant A | 79.2 (2.8) | 85.9 (2.5)
  Participant B: number analyzed (Participants) | 1 | 1
  Participant B | 61.8 (11.4) | 49.0 (2.3)
  Participant C: number analyzed (Participants) | 1 | 1
  Participant C | 87.0 (3.6) | 95.8 (2.6)
Statistical Analysis 1: Comparison: SIT With Habitual Prosthesis vs STAND With Habitual Prosthesis; Test type: Other; [other analysis details as in outcome 1, analysis 1]

8. Secondary Outcome: Percentage of Body Weight on Contralateral Limb at 65 Degrees Knee Flexion
Description: as for outcome 7
Time Frame: as for outcome 2
Population: Each participant served as their own control in this analysis.
Measure: Mean (Standard Deviation); unit: % body weight
Groups:
- SIT With Assist-Knee (Settings 1): Contralateral limb weight distribution during stand-to-sit at 65 degrees knee flexion when using Assist-Knee (Settings 1).
- STAND With Assist-Knee (Settings 1): Contralateral limb weight distribution during sit-to-stand at 65 degrees knee flexion when using Assist-Knee (Settings 1).
- SIT With Assist-Knee (Settings 2): Contralateral limb weight distribution during stand-to-sit at 65 degrees knee flexion when using Assist-Knee (Settings 2).
- STAND With Assist-Knee (Settings 2): Contralateral limb weight distribution during sit-to-stand at 65 degrees knee flexion when using Assist-Knee (Settings 2).
Arm/Group | SIT With Assist-Knee (Settings 1) | STAND With Assist-Knee (Settings 1) | SIT With Assist-Knee (Settings 2) | STAND With Assist-Knee (Settings 2)
Number analyzed (Participants) | 3 | 3 | 3 | 3
% body weight
  Participant A: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant A | 67.7 (7.5) | 82.0 (1.9) | 48.0 (9.4) | 83.5 (1.2)
  Participant B: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant B | 23.5 (13.7) | 27.0 (6.9) | 19.4 (10.4) | 31.3 (2.3)
  Participant C: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant C | 67.0 (1.6) | 78.6 (4.5) | 63.4 (9.9) | 76.4 (3.2)
Statistical Analysis 1: Comparison: SIT With Assist-Knee (Settings 1) vs STAND With Assist-Knee (Settings 1) vs SIT With Assist-Knee (Settings 2) vs STAND With Assist-Knee (Settings 2); Test type: Other; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the experimental sessions with each participant, up to 3 hours.
Arm/Group | Study Participants
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
This clinical trial collected data with a small number of participants. These results may not be generalizable to the entire population. Furthermore, this clinical trial used the Assist-Knee experimental prototype which is in a proof-of-concept stage. There is a potential for the outcome measures to improve as the Assist-Knee device design is refined through development.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT04023045/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT04023045/SAP_001.pdf